CLINICAL TRIAL: NCT06966648
Title: Effect of Core Stabilization Training on Balance and Pivot Performance in Young Rhythmic Gymnasts: A Pilot Randomized Controlled Trial
Brief Title: Pilot Study on Core Stabilization Training on Stable vs Unstable Surfaces in Young Rhythmic Gymnasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Assistant Professor, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-11 2025
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Postural Balance; Motor Skills; Physical Fitness; Athletic Performance
Keywords: Rhythmic gymnastics; Core stabilization; Balance training; Unstable surfaces; Pilot trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stable Surface Group (Active Comparator): Participants will perform a core stabilization program on stable surfaces (e.g., floor, foam blocks). Exercises target trunk control and balanc
  Interventions: Other: Core stabilization on stable surfaces
- Unstable Surface Group (Experimental): Participants will perform the same core stabilization program on unstable surfaces (e.g., BOSU, wobble board).
  Interventions: Other: Core stabilization on unstable surfaces

INTERVENTIONS:
Other: Core stabilization on stable surfaces — Participants will perform a structured core stabilization training program on stable surfaces, such as the floor and rigid foam blocks. The program includes functional exercises targeting trunk control, postural alignment, and balance, delivered three times per week over a 7-week period.
  Arms: Stable Surface Group
Other: Core stabilization on unstable surfaces — Participants will perform the same structured core stabilization training program as the stable surface group, but on unstable surfaces such as BOSU balls and wobble boards. The intervention is designed to challenge balance, proprioception, and core muscle activation. Sessions are conducted three times per week over a 7-week period.
  Arms: Unstable Surface Group

SUMMARY:
This pilot randomized controlled trial will investigate the effects of a 7-week core stabilization program performed on stable versus unstable surfaces in young competitive rhythmic gymnasts. Sixteen athletes will be randomized into two groups and will be assessed for changes in static balance and pivot performance.

DETAILED DESCRIPTION:
Rhythmic gymnastics requires high-level neuromuscular control, especially for skills involving balance and rotation. Core stabilization exercises are commonly included in training, but limited evidence exists regarding the impact of surface type on training effectiveness. This pilot study will compare the effects of a 7-week core stabilization program conducted on stable versus unstable surfaces on balance and pivot execution in rhythmic gymnasts aged 7-12. Participants will be randomly allocated into two equal groups and will be assessed pre- and post-intervention on selected balance and pivot tasks in accordance with Fédération Internationale de Gymnastique (FIG) standards. The study aims to inform future trials by estimating effect sizes and assessing the feasibility of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Female rhythmic gymnasts aged 7 to 12 years
* Minimum of 1 year of experience in rhythmic gymnastics
* Active participation in organized training at least 3 times per week
* No current musculoskeletal pain or injury
* Ability to perform all training and assessment tasks safely
* Written informed consent provided by a parent or legal guardian

Exclusion Criteria:

* History of acute lower limb or spinal injury within the past 6 months
* Presence of neurological, orthopedic, or vestibular disorders affecting balance
* Concurrent participation in other structured physical training programs outside rhythmic gymnastics
* Any medical condition that would contraindicate participation in physical exercise

Ages: 7 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Balance Duration | Baseline and Week 7 (post-intervention)
  Balance performance will be measured in seconds using a handheld stopwatch (Ultrak 250 Stopwatch Chronometer). Each gymnast will perform three static balance elements (passé, attitude, and side split with help) in relevé position while wearing half shoes. The timer will start once the gymnast achieves final posture and stop when balance is lost, form deteriorates, or the center of gravity shifts. Five trials will be performed for each element, and the longest successful attempt will be recorded. All tests will be performed with eyes open.
Pivot Performance (Number of Clean Rotations) | Baseline and Week 7 (post-intervention)
  Pivot performance will be assessed as the number of clean, full rotations executed without technical faults, based on Fédération Internationale de Gymnastique (FIG) regulations. Each gymnast will perform two pivot elements (passé forward and attitude) in relevé position while wearing half shoes, maintaining proper form and control. Five attempts will be performed for each pivot type, and the highest number of clean rotations will be recorded. All tests will be performed with eyes open.

CONTACTS AND LOCATIONS:
Locations (1):
- International Hellenic University, Thessaloniki, Greece, Greece